CLINICAL TRIAL: NCT03187184
Title: Implementing Preemptive Pharmacogenomic Testing for Colorectal Cancer Patients in a Community Oncology Clinic
Acronym: CRCPGx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essentia Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 021870
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single arm proof of concept trial. Sequential boundaries will be used to monitor late PGx test returns (failure to receive OneOme RightMed® pharmacogenomic test results before initiating chemotherapy). The concept will be considered a failure if excessive numbers of late PGx test returns are seen, that is, if the number of late PGx test returns is equal to or exceeds bn out of n patients (see table below). This Pocock-boundary is based upon the probability of early failure when the rate of late PGx test returns is equal to the acceptable rate [event probability θ]. In this trial crossing the boundary will not result in early stopping, because chemotherapy treatment is not dependent upon receipt of PGx test results prior to treatment initiation, but may be used to revise future protocol methodology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OneOme RightMed® Test (Experimental): OneOme RightMed® currently tests for 22 genes that impact over 340 drugs used in multiple fields of medicine, including oncology. The drugs tested for by OneOme RightMed® were generated from practice guidelines and the FDA's guidelines for genotyping, and drugs with published, clinical evidence supporting genotyping. Testing is done using a prepackaged OneOme RightMed® kit to collect a buccal swab. OneOme RightMed® PGx test uses a DNA Genotek ORAcollect OC-100 buccal swab kit to extract DNA, which is then analyzed through polymerase chain reaction (PCR).
  Interventions: Device: OneOme RightMed®

INTERVENTIONS:
Device: OneOme RightMed® — OneOme RightMed® currently tests for 22 genes that impact over 340 drugs used in multiple fields of medicine, including oncology. The drugs tested for by OneOme RightMed® were generated from practice guidelines and the FDA's guidelines for genotyping, and drugs with published, clinical evidence supporting genotyping. Testing is done using a prepackaged OneOme RightMed® kit to collect a buccal swab. OneOme RightMed® PGx test uses a DNA Genotek ORAcollect OC-100 buccal swab kit to extract DNA, which is then analyzed through polymerase chain reaction (PCR).

SUMMARY:
Pharmacogenomics (PGx) studies the interactions between an individuals genes and medications. PGx testing identifies genes within an individual that may affect treatment, efficacy, and toxicity of drugs. With improvements in testing speed, accuracy and cost, it is now possible to perform PGx testing in cancer patients prior to starting chemotherapy. The test results may help a physician personalize chemotherapy dosing. The goal of this study is to determine if PGx testing using the OneOme® Rightmed test is feasible in a community oncology clinic to guide treatment prior to starting chemotherapy. The study will also gather data regarding the frequency of genes within the local population as well as the impact of testing on chemotherapy doses.

DETAILED DESCRIPTION:
The goal of personalized medicine is to tailor therapies to an individual patient with a goal of maximizing benefit and minimizing treatment related side effects. Inter-individual variability in metabolic enzymes can have a significant impact on cancer therapies. Pharmacogenomics (PGx) studies the interactions between drugs and genes, and pharmacogenomic screening tests can assess for genetic variations among individuals to personalize medicine. PGx testing identifies genes within an individual that may affect treatment, efficacy, and toxicity of drugs. PGx screening prior to chemotherapy would help identify patients with genetic polymorphisms that are at increased risk for drug toxicity and would benefit from genetic-guided dosing, resulting in decreased risk of adverse events (AEs) related to the chemotherapy. PGx testing is not routinely used in community-based oncology practices. The cost of testing as well as lengthy waits for results have limited routine use of this testing. Advances in testing have reached the point where routine preemptive testing could benefit patients with newly diagnosed cancer.

PGx testing evaluating a large number of metabolic enzymes is now commercially available. OneOme RightMed® is a privately owned company developed by doctors and scientists at Mayo Clinic with a mission "to provide the most cost-effective, comprehensive, personalized, pharmacogenomics analysis integrated into everyday clinical care." OneOme RightMed® currently tests for 22 genes that impact over 340 drugs used in multiple fields of medicine, including oncology. The drugs tested for by OneOme RightMed® were generated from practice guidelines and the FDA's guidelines for genotyping, and drugs with published, clinical evidence supporting genotyping. With developments in sequencing technology, comprehensive PGx testing can now be completed for a modest cost. Testing is done using a prepackaged OneOme RightMed® kit to collect a buccal swab. OneOme RightMed® PGx test uses a DNA Genotek ORAcollect OC-100 buccal swab kit to extract DNA, which is then analyzed through polymerase chain reaction (PCR). The results are available in 10 or less calendar days to the provider and/or pharmacist. The report provides "genotype-derived recommendations" with additional quick references for medication dosing guidance.

Despite clear clinical implications, incorporation of PGx testing has historically been challenging due to potential delay in initiation of therapy and uncertainty of clinical and economic benefits. However, in the past decades, clinically actionable gene-drug interactions, such as the polymorphisms discussed above, have been identified. Additionally, the availability of high-quality genotyping in a timely manner with lower costs makes PGx testing feasible. Pilot studies implementing PGx testing have been conducted at academic centers.10,13-15 Though the knowledge gained from those studies enhanced their ability to implement PGx testing, pilot studies implementing PGx testing in a community-based health care setting in oncology treatment have not been conducted, to the best of our knowledge. Therefore, our pilot study would evaluate the feasibility of implementing PGx testing in routine oncology treatment at a community-based health care center. CRC is a common cancer and the drugs used in treating CRC are affected by PGx. Thus, CRC represents an ideal situation to evaluate the feasibility of routine preemptive PGx testing. While this study represents an initial pilot feasibility study, our ultimate goal is to evaluate the benefits of PGx in the community setting in regards to reduction of toxicity, improved cancer outcomes, and cost savings.

Primary Objective

1. To determine if preemptive PGx testing is feasible in a community oncology clinic.

Secondary Objective

1. To gather pilot data on the proportion of Essentia Health patients with metabolic enzyme alleles that could impact chemotherapy dosing.
2. To evaluate the impact of PGx guided chemotherapy dosing on toxicity.
3. To evaluate the cost-effectiveness of PGx testing in Essentia Health patients with colorectal cancer.

Eligible patients will have a histological diagnosis of colorectal cancer. The intent of the study is to enroll patients as quickly as possible once a decision has been made that a patient is a candidate for chemotherapy for stage 2-4 colorectal cancer. While many patients will be eligible for study participation at their initial consultation with medical oncology, it is also anticipated that some patients may need additional testing prior to eligibility. This would also include patients who have been followed in the medical oncology department that develop a new malignancy or have a recurrence. Patients must be enrolled to the study within 7 days of their initial consultation, or within 7 days of a physician visit, after any additional tests or biopsies have been completed, when the patient is felt to be a suitable candidate for chemotherapy. After obtaining informed consent from eligible patients, a commercially available pharmacogenomics panel, the OneOme RightMed® pharmacogenomic test, will be ordered. Patients will not be responsible for the cost of PGx testing. The study will not prescribe any specific chemotherapy regimens. All decisions regarding the clinical care of the patient will be made by the treating physician. Treatment will not be delayed to wait for PGx results per study protocol, however the treating physician may elect to do so. When PGx test results are available, results will be interpreted by the Oncology Lead Pharmacist at Essentia Health, and recommendations will be made to the treating physician regarding potential chemotherapy does adjustments. The treating physician will have the ultimate decision as to whether chemotherapy dose adjustments are done as a result of PGx testing. Patients will be seen by study staff prior to initiating chemotherapy, and after chemotherapy cycles 1-3 to assess for toxicity and to determine if any dose modifications were done by the treating physician.

Patient demographic data will be collected at baseline. Once patients start chemotherapy, treatment toxicity data will be collected prior to chemotherapy and after cycles 1-3. For patients receiving continuous chemotherapy such as infusional 5-FU or capecitabine concurrent with radiation, a cycle will be defined as 2 weeks. Toxicity data will be collected following Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Data will be collected for common side effects associated with typical colorectal cancer chemotherapy regimens including, leukopenia, neutropenia, anemia, thrombocytopenia, fatigue, nausea/vomiting, diarrhea, mucositis, hand-foot syndrome, peripheral neuropathy, and abdominal pain. Other toxicities identified by study staff will be collected as well. Chemotherapy dose modifications made by the treating physician will be collected for chemotherapy cycles 1-3.

When PGx results are available, study staff will alert the Oncology Lead Pharmacist who will evaluate the results and make recommendations to the treating physician regarding suggested dose modification to the planned chemotherapy regimen. The primary assessment of the analysis will focus on UGT1A1 and DPD.

In cases where the suggested dose modifications are unclear or the results are atypical, the Lead Pharmacist will consult with OneOme RightMed® staff to determine appropriate recommendations. The Lead Pharmacist will also review each patient's current medication list and identify if there are any additional medication concerns related to evaluated genes other than UGT1A1 and DPYD. Any identified additional concerns will be noted on the Results Interpretation and Impact form. Once the form is complete, a copy will be forwarded to the treating physician who will then complete the form to indicate whether any changes to the planned chemotherapy regimen will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven Stage 2-4 colon or rectal adenocarcinoma with an anticipated need for chemotherapy, which may include neoadjuvant, adjuvant or palliative treatment, and may include oral or intravenous chemotherapy.
2. Adequate organ function and performance status to receive chemotherapy as determined by the treating physician.
3. Age ≥ 18 years.
4. Ability to understand and the willingness to sign a written informed consent documented.
5. Patients must sign consent within 7 days of the physician visit for newly diagnosed or recurrent colorectal cancer when a patient is initially felt to be a candidate for chemotherapy.

Exclusion Criteria:

1. Patients received prior chemotherapy for colorectal cancer in the last 12 months.
2. Patients received prior OneOme RightMed® pharmacogenomic testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
PGx Test Interpretation | 10 days
  Proportion of patients with pharmacogenomic testing completed and interpreted prior to starting chemotherapy.

SECONDARY OUTCOMES:
Allele Frequency | 10 days
  The proportion of Essentia Health patients with metabolic enzyme alleles that could impact chemotherapy dosing will be reported. Descriptive statistics, proportion and 95% confidence interval (95% CI), will be reported.
Chemotherapy Toxicity | 3 months
  Toxicity will be reported for all patients and the sub-groups of patients with and without the metabolic enzyme alleles that could impact chemotherapy. Descriptive statistics, proportion and 95% confidence interval (95% CI), will be reported. Depending upon the sample sizes involved, either the chi-square test or Fisher's exact test will be used to compare the sub-groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Friday, MD, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No